CLINICAL TRIAL: NCT00267969
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo Controlled Trial Evaluating the Efficacy and Safety of Ustekinumab (CNTO 1275) in the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study of Safety and Effectiveness of Ustekinumab (CNTO 1275) in Patients With Moderate to Severe Plaque-type Psoriasis
Acronym: PHOENIX1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor Research & Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006328; C0743T08 (Other: Centocor Research & Development, Inc., PA, USA); 2005-003529-15 (EudraCT Number); NCT01585714 (obsolete NCT alias)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Psoriasis
Keywords: Ustekinumab; CNTO1275; Plaque type Psoriasis; Interleukin-23; IL-23; Psoriasis; Interleukin 12; IL-12
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ustekinumab 45 mg (Experimental): Patients received ustekinumab 45 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 40, patients who achieved PASI 75 at both Week 28 and Week 40 were re-randomized to withdraw from therapy (placebo) or continue 45 mg every 12 week maintenance therapy.
  Interventions: Drug: ustekinumab
- ustekinumab 90 mg (Experimental): Patients received ustekinumab 90 mg at Week 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 40, patients who achieved PASI 75 at both Week 28 and Week 40 were re-randomized to withdraw from therapy (placebo) or continue 90 mg every 12 week maintenance therapy.
  Interventions: Drug: ustekinumab
- Placebo (Placebo Comparator): Patients received placebo at Weeks 0 and 4. At Weeks 12 and 16, placebo crossed over to receive ustekinumab 45 mg or 90 mg. Treatments after Week 16 were dependent on clinical response.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ustekinumab — Type = exact number, Form = solution for injection, Number = 45 and 90, Unit = mg, Route = subcutaneous (SC) administered at Weeks 0, 4 and 16. Both treatments (45 mg and 90 mg) administered every 12 weeks after Week 16 depending on clinical response.
  Other Names: CNTO 1275
  Arms: ustekinumab 45 mg; ustekinumab 90 mg
Drug: placebo — Form = solution for injection, route = SC administered at Weeks 0 and 4. At Weeks 12 and 16, placebo will be crossed over to receive ustekinumab 45 mg or 90 mg.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness and safety of ustekinumab (CNTO 1275) in the treatment of patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized (patients are assigned to different treatments based on chance), double blind (neither the patient nor the physician knows whether medication or placebo [an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study] is being taken, or at what dosage), parallel-group (each group of patients are treated at the same time), multicenter study to determine the effectiveness and safety of two different doses of ustekinumab administered subcutaneously (under the skin) as compared with placebo in patients with moderate to severe plaque-type psoriasis (the most common type of psoriasis). 766 patients will be randomized to Group 1 (ustekinumab 45 mg), Group 2 (ustekinumab 90 mg) and Group 3 (placebo) at Week 0. The study was designed to evaluate the effectiveness and safety of 2 dose regimens of ustekinumab: (1) 45 mg at Weeks 0 and 4 followed by 45 mg every 12 weeks maintenance therapy (treatment designed to help the original primary treatment succeed) and (2) 90 mg at Weeks 0 and 4 followed by 90 mg every 12 weeks maintenance therapy. The study will consist of 4 periods: (1) Placebo-controlled portion of study [Week 0 to Week 12] during which the safety and effectiveness of 2 doses (45mg and 90mg) of ustekinumab will be compared to placebo; (2) Placebo crossover and active treatment portion of study [Week 12 to Week 40] during which patients randomized to receive placebo at Week 0 will crossover to receive ustekinumab, and all patients will receive active treatment; (3) Randomized withdrawal portion of study [beginning at Week 40] during which patients who received ustekinumab [45mg or 90mg every 12 weeks] at Week 0 and are responding to it, will be randomized either to placebo or continued maintenance therapy with ustekinumab; and (4) Long-term extension [from Week 52 to Week 264 (ie, 5 years)] period during which the safety and effectiveness of ustekinumab long-term use will be evaluated in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plaque-type psoriasis diagnosed at least 6 months prior and covering at least 10% of total body surface areas
* Have psoriasis area-and-severity index score of >=12
* Patients who are considered by treating dermatologist to be a candidate for phototherapy or systemic treatment of psoriasis
* Have no history of latent or active TB

Exclusion Criteria:

* Currently have nonplaque forms of psoriasis or drug-induced psoriasis
* Have any therapeutic agent targeted at reducing IL-12 or IL-23
* Have had a BCG vaccination within the previous 12 months
* Have a history of chronic or recurrent infectious disease or who have or have had a serious infection requiring hospitalization or intravenous antibiotics within the previous 2 months
* Have or ever have had a nontuberculous mycobacterial infection or opportunistic infection
* Patients known to be infected with human immunodeficiency virus, hepatitis B, or hepatitis C
* Have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Patients with a malignancy or who have a history of malignancy (with the exception of certain skin cancers and pre-invasive cervical cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Research & Development, Inc. Clinical Trial, Study Director — Centocor Research & Development, Inc.
Locations (42):
- United States (28):
  - Phoenix, Arizona
  - Los Angeles, California
  - Redwood City, California
  - Santa Monica, California
  - Denver, Colorado
  - Wilmington, Delaware
  - Ocala, Florida
  - Alpharetta, Georgia
  - Marietta, Georgia
  - Newnan, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Normal, Illinois
  - Indianapolis, Indiana
  - Lake Charles, Louisiana
  - Worcester, Massachusetts
  - Fridley, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - East Windsor, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Goodlettsville, Tennessee
  - Dallas, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Belgium (2):
  - Brussels
  - Edegem
- Canada (12):
  - Edmonton, Alberta
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - London, Ontario
  - North Bay, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec

REFERENCES:
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Leonardi CL, Kimball AB, Papp KA, Yeilding N, Guzzo C, Wang Y, Li S, Dooley LT, Gordon KB; PHOENIX 1 study investigators. Efficacy and safety of ustekinumab, a human interleukin-12/23 monoclonal antibody, in patients with psoriasis: 76-week results from a randomised, double-blind, placebo-controlled trial (PHOENIX 1). Lancet. 2008 May 17;371(9625):1665-74. doi: 10.1016/S0140-6736(08)60725-4. PMID 18486739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, 766 patients were randomized in North America and Europe to receive either placebo or ustekinumab (CNTO 1275).
Groups:
- Placebo (CP): Controlled period (Week 0-12) - Placebo group
- Ustekinumab 45 mg (CP): Controlled period (Week 0-12) - Ustekinumab 45 mg group
- Ustekinumab 90 mg (CP): Controlled period (Week 0-12) - Ustekinumab 90 mg group
- Placebo -> Ustekinumab 45 mg (After CP): After Controlled period (Week 12-264) - patients receiving Placebo at Weeks 0 and 4 -> receiving ustekinumab 45 mg every 12 weeks (q12wk) or every 8 weeks (q8wk) from Week 12 to Week 244. Some patients were withdrawn from ustekinumab at Week 40 and re-treated with ustekinumab 45 q12w.
- Placebo -> Ustekinumab 90 mg (After CP): After Controlled period (Week 12-264) - patients receiving Placebo at Weeks 0 and 4 -> receiving ustekinumab 90 mg q12wk or q8wk from Week 12 to Week 244. Some patients were withdrawn from ustekinumab at Week 40 and re-treated with ustekinumab 90 q12w.
- Ustekinumab 45 mg (After CP): After Controlled period (Week 12-264) - patients receiving ustekinumab 45 mg at Weeks 0 and 4 -> receiving ustekinumab 45 mg q12wk or q8wk from Week 16 to Week 244. Some patients were withdrawn from ustekinumab at Week 40 and re-treated with ustekinumab 45 q12w.
- Ustekinumab 90 mg (After CP): After Controlled period (Week 12-264) - patients receiving ustekinumab 90 mg at Weeks 0 and 4 -> receiving ustekinumab 90 mg q12wk or q8wk from Week 16 to Week 244. Some patients were withdrawn from ustekinumab at Week 40 and re-treated with ustekinumab 90 q12w.
Period: Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 255 (Number of patients randomized) | 255 (Number of patients randomized) | 256 (Number of patients randomized) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to Controlled Period.)
Completed | 243 | 254 | 245 | 0 | 0 | 0 | 0
Not Completed | 12 | 1 | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 6 | 0 | 0 | 0 | 0
Period: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Controlled Period.) | 123 | 120 | 254 | 245
Completed | 0 | 0 | 0 | 87 | 85 | 172 | 173
Not Completed | 0 | 0 | 0 | 36 | 35 | 82 | 72
Not completed — Adverse Event | 0 | 0 | 0 | 7 | 8 | 23 | 21
Not completed — Death | 0 | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 10 | 6 | 28 | 15
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5 | 8 | 9 | 10
Not completed — Other | 0 | 0 | 0 | 13 | 11 | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg | Total
Number analyzed (Participants) | 255 | 255 | 256 | 766
Age Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (11.32) | 44.8 (12.48) | 46.2 (11.27) | 45.3 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 80 | 83 | 235
  Male | 183 | 175 | 173 | 531

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area-and-severity Index (PASI) 75% Improvement From Baseline at Week 12.
Description: The number of participants achieving at least 75% improvement from baseline in Psoriasis Area and Severity Index (PASI) (0 [best] - 72 [worst]) at Week 12. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: Week 12
Population: Intent to treat. All patients randomized were included in the analysis according to the assigned treatment groups. Patient is considered a non- responder if the patient has used any pre-specified prohibited medications or discontinued due to lack of efficacy, or an AE of worsening of psoriasis, or had missing data at Week 12.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 255 | 255 | 256
Participants | 8 | 171 | 170
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and placebo at an overall significance level of 0.05. Sample Size: With 750 patients (250 in each treatment group), simulation studies were conducted to calculate the power to detect a treatment difference in the primary endpoint between ustekinumab groups and placebo using a CMH test stratified by baseline weight [<=90kg vs > 90 kg). For all the scenarios evaluated, the power is >99% at an overall significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square — To control for the multiplicity for the primary endpoint analysis, the Holm's procedure was used at an overall significance level of 0.05; Stratified by baseline weight [≤ 90kg vs > 90 kg)]

2. Secondary Outcome: Number of Participants Who Achieved a Physician Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 12
Description: The PGA is used to determine the participant's psoriasis lesions overall at a given time point. Overall lesions will be graded as : (0) = cleared, (1) = minimal, (2) = mild, (3) = moderate, (4) = marked, and (5) = severe for induration, erythema, and scaling. The sum of the 3 scales will be divided by 3 to obtain a final PGA score ranging from 0 [best] to 5 [worst].
Time Frame: Week 12
Population: Intent to treat. All patients were included in the analysis according to the assigned treatment groups. Patient is considered a non- responder if the patient has used any pre-specified prohibited medications or discontinued due to lack of efficacy, or an AE of worsening of psoriasis, or had missing data at Week 12.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 255 | 255 | 256
participants | 10 | 151 | 156
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel(CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and placebo at an overall significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square — To control the multiplicity for the primary and the secondary endpoint analyses, Holm's procedure was used but the two comparisons for the primary endpoint and the two comparisons for the 1st second endpoint analyses need to be significant first; Stratified by baseline weight [≤ 90kg vs > 90 kg)]

3. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 12
Description: Change from baseline in Dermatology Life Quality Index (DLQI) from baseline at Week 12. This DLQI is a 10-item questionnaire, that in addition to evaluating overall quality of life, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Scores range from 0 (no impairment in quality of life) to 30 (most impairment in quality of life).
Time Frame: Baseline (Week 0), Week 12
Population: Patients were included in the analysis according to the assigned treatment groups. Zero change is imputed if the patient has used any pre-specified prohibited medications or discontinued due to lack of efficacy. Other missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Placebo | Ustekinumab 45 mg | Ustekinumab 90 mg
Number analyzed (Participants) | 252 | 254 | 249
Scores on a scale | 0.0 [-3.0 to 3.0] | -6.0 [-12.0 to -3.0] | -7.0 [-12.0 to -4.0]
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; Treatment and patient's baseline weight (≤ 90kg vs > 90 kg) as factors in the model
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and placebo at an overall significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores — [p-value comment as in outcome 2, analysis 2]; Treatment and patient's baseline weight (≤ 90kg vs > 90 kg) as factors in the model

4. Secondary Outcome: Psoriasis Area and Severity Index (PASI) 75 Responders at Week 52
Description: The number of participants achieving at least 75% improvement from baseline in Psoriasis Area and Severity Index (PASI) (0 [best] - 72 [worst]) at Week 52 in participants randomly assigned to a treatment group at Week 40. This is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: Week 52
Population: Patients were included in the analysis according to the assigned treatment groups. Patient is considered a non- responder if the patient has used any pre-specified prohibited medications or discontinued due to lack of efficacy. Other missing data were not imputed.
Measure: Number; unit: participants
Groups:
- Group 1: Ustekinumab 45 mg Withdrawal Group: Patients received ustekinumab 45 mg at Weeks 0, 4, 16 and 28.
- Group 2: Ustekinumab 45 mg Every 12 Weeks: Patients received ustekinumab 45 mg at Weeks 0, 4, 16, 28 and 40.
- Group 3: Ustekinumab 90 mg Withdrawal: Patients received ustekinumab 90 mg at Weeks 0, 4, 16 and 28.
- Group 4: Ustekinumab 90 mg Every 12 Weeks: Patients received ustekinumab 90 mg at Weeks 0, 4, 16, 28 and 40.
- Group 5: Withdrawal Combined Group: Groups 1 and 3 (Withdrawal Combined)
- Group 6: Combined Ustekinumab Every 12 Weeks: Groups 2 and 4 (Combined Ustekinumab every 12 weeks)
Arm/Group | Group 1: Ustekinumab 45 mg Withdrawal Group | Group 2: Ustekinumab 45 mg Every 12 Weeks | Group 3: Ustekinumab 90 mg Withdrawal | Group 4: Ustekinumab 90 mg Every 12 Weeks | Group 5: Withdrawal Combined Group | Group 6: Combined Ustekinumab Every 12 Weeks
Number analyzed (Participants) | 73 | 77 | 86 | 85 | 159 | 162
participants | 47 | 67 | 53 | 77 | 100 | 144
Statistical Analysis 1: Comparison: Group 5: Withdrawal Combined Group vs Group 6: Combined Ustekinumab Every 12 Weeks; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 2: Comparison: Group 3: Ustekinumab 90 mg Withdrawal vs Group 4: Ustekinumab 90 mg Every 12 Weeks; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [≤ 90kg vs > 90 kg)]
Statistical Analysis 3: Comparison: Group 1: Ustekinumab 45 mg Withdrawal Group vs Group 2: Ustekinumab 45 mg Every 12 Weeks; Null Hypothesis: No difference between combined maintenance group and the combined withdrawal group, ustekinumab 90 mg maintenance group and the withdrawal group, ustekinumab 45 mg maintenance group and the withdrawal group at an overall significance level of 0.05; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel (CMH) chi square — To control the overall multiplicity, the combined groups was tested first and each dose will then be tested; but the primary and the 1st 2 secondary endpoint analyses need to be significant before this endpoint can be tested; Stratified by baseline weight [≤ 90kg vs > 90 kg)]

ADVERSE EVENTS:
Time Frame: 264 weeks
Description: In adverse events reporting: 1 patient not included was randomized in Ustekinumab 90 mg Controlled period (CP) but not treated. 1 patient included in Ustekinumab 45 mg (after CP) and 6 patients included in Ustekinumab 90 mg (after CP) had discontinued study agent during the CP but had follow-up after CP.
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 2/255 | 2/255 | 4/255 | 20/123 | 18/120 | 38/255 | 33/251
Other Adverse Events (participants affected / at risk) | 81/255 | 102/255 | 84/255 | 110/123 | 102/120 | 207/255 | 207/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=255) | Ustekinumab 45 mg (CP) (N=255) | Ustekinumab 90 mg (CP) (N=255) | Placebo -> Ustekinumab 45 mg (After CP) (N=123) | Placebo -> Ustekinumab 90 mg (After CP) (N=120) | Ustekinumab 45 mg (After CP) (N=255) | Ustekinumab 90 mg (After CP) (N=251)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 3
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Asymptomatic HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chorea (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Renal infarct (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=255) | Ustekinumab 45 mg (CP) (N=255) | Ustekinumab 90 mg (CP) (N=255) | Placebo -> Ustekinumab 45 mg (After CP) (N=123) | Placebo -> Ustekinumab 90 mg (After CP) (N=120) | Ustekinumab 45 mg (After CP) (N=255) | Ustekinumab 90 mg (After CP) (N=251)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 3 | 13 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 2 | 5 | 9 | 18 | 18
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 1 | 4 | 2 | 13 | 4
Nausea (Gastrointestinal disorders) | 3 | 4 | 2 | 7 | 3 | 12 | 10
Fatigue (General disorders) | 3 | 5 | 6 | 9 | 5 | 8 | 5
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 11 | 16 | 25 | 29
Cellulitis (Infections and infestations) | 2 | 2 | 0 | 1 | 6 | 7 | 5
Gastroenteritis (Infections and infestations) | 5 | 6 | 2 | 11 | 11 | 23 | 25
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 1 | 1 | 6 | 12 | 7
Influenza (Infections and infestations) | 3 | 3 | 2 | 16 | 15 | 28 | 27
Nasopharyngitis (Infections and infestations) | 22 | 26 | 21 | 47 | 36 | 70 | 75
Pharyngitis (Infections and infestations) | 3 | 2 | 1 | 9 | 6 | 11 | 12
Sinusitis (Infections and infestations) | 6 | 6 | 4 | 15 | 14 | 37 | 31
Tooth abscess (Infections and infestations) | 0 | 1 | 2 | 5 | 7 | 16 | 13
Upper respiratory tract infection (Infections and infestations) | 16 | 18 | 16 | 43 | 34 | 82 | 77
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 3 | 6 | 14 | 9
Viral upper respiratory tract infection (Infections and infestations) | 1 | 4 | 3 | 5 | 10 | 19 | 14
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 7 | 4 | 14 | 15
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 11 | 9 | 22 | 17
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 13 | 14 | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 10 | 6 | 10 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 6 | 20 | 13 | 31 | 33
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 4 | 7 | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 7 | 13 | 18 | 23 | 27
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7 | 10 | 7 | 15
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 9 | 2 | 16 | 7
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 6 | 5 | 2
Headache (Nervous system disorders) | 6 | 14 | 13 | 15 | 7 | 24 | 17
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 4 | 6 | 16 | 7
Depression (Psychiatric disorders) | 3 | 5 | 2 | 7 | 6 | 8 | 12
Insomnia (Psychiatric disorders) | 2 | 2 | 2 | 7 | 7 | 12 | 14
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 6 | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 13 | 7 | 13 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 10 | 8 | 3 | 13
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 13 | 5 | 11 | 11
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 7 | 2 | 6 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 7 | 6 | 7 | 7
Hypertension (Vascular disorders) | 4 | 5 | 3 | 14 | 17 | 21 | 30
Upper respiratory tract infection (Infections and infestations) | 16 | 18 | 16 | 43 | 34 | 82 | 77

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse event (NAE) excludes patients who only had NAE that occured in <=5% of patients. This information may vary from existing approved labeling and publications due to the requirements of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.